CLINICAL TRIAL: NCT04362631
Title: Advanced, Bio-Integrated, and Cloud-Enabled Sensors for Early Diagnosis of Respiratory Infections in the Home Setting
Brief Title: Respiratory Infection Monitoring
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ankit Bharat, Principal Investigator, Northwestern University
Other Study IDs: STU00210701
Record Dates: First submitted 2020-03-30; First posted 2020-04-27 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Adults 18 years or older

SUMMARY:
This study will monitor physical bio-markers such as heart rate, respiratory rate, and temperature to detect potential respiratory infections.

DETAILED DESCRIPTION:
The advanced, bio-integrated wireless sensor (ADAM) that provides a comprehensive assessment of cardiopulmonary health. The technology employs advanced low-power operation, in-sensor analytics, and cloud integration. The sensor's novel soft mechanics allows for comfortable placement on the suprasternal notch, a location of unique anatomical importance, to collect both core vitals (heart rate, respiratory rate, temperature, and physical activity including sleep quality) and novel respiratory digital biomarkers (cough count, swallowing, throat clearing and respiratory effort). The investigators will deploy this system in a cohort of high-risk patients for respiratory infection in a home setting to predict for respiratory infections prior to clinical deterioration.

The investigators aim to capture data on 122 study subjects over the course of 52 weeks of continuous wear or the investigator's device to thoroughly characterize physiological data and diagnosis of respiratory infections. Data from standard of care appointments, diagnostic testing or imaging, or treatment will be collected from the patient medical record to validate device data.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Outpatient at start of the study
* Established clinical history of COPD
* Previous hospital or ICU admission for pneumonia or COPD
* Active corticosteroid prescription
* Willingness to participate in the study (long term continuous wear of the device)
* Ability to apply and remove devices and use a mobile application

Exclusion Criteria:

* Mental or neurodegenerative disease
* Including a current diagnosis of asthma, respiratory disorders (e.g. active tuberculosis, lung cancer, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases); pneumonia or other RTIs not resolved ≤14 days or ≤7 days, respectively, prior to screening
* Skin condition or wound on suprasternal notch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of wearable device to detect respiratory infection parameters: cough count | 1 year
  Device data measuring cough count. Captured by analysis of peak acclerometer graphing and duration in meters per second squared (m/s2).
Monitoring of respiratory infection symptoms, WURSS-11 Survey | 1 year
  WURSS-11 survey. https://www.fammed.wisc.edu/files/webfm-uploads/documents/research/wurss-11.pdf The WURSS-11 survey will be conducted on a weekly basis by study subjects for the duration of the study (up to 52 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No